CLINICAL TRIAL: NCT04773340
Title: Adapting Dialectical Behavior Therapy for the Treatment of Criminal Offenders With Antisocial Personality Disorder
Acronym: DBT-ASPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fordham University (Other)
Responsible Party: Principal Investigator, Barry Rosenfeld, Professor/Principle Investigator, Fordham University
Other Study IDs: 957186
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Antisocial Personality Disorder
MeSH Terms: conditions — Antisocial Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DBT intervention: Adaptation of Dialectical Behavior Therapy designed for repeat criminal offenders at high risk of reoffense.
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Behaviorally-focused intervention for individuals with personality disorder and a history of significant behavioral problems.

SUMMARY:
This pilot study is intended to adapt and refine an intervention grounded in the principles of Dialectical Behavior Therapy, for the treatment of repeat criminal offenders with antisocial personality disorder. This study will be open to individuals participating in an intensive supervision program operated by the U.S. District Court of the Southern District of New York (the RISE Court program).

DETAILED DESCRIPTION:
Antisocial personality disorder (ASPD) is among the most damaging and costly mental disorders, yet little research has sought to address the root causes of this disorder. Indeed, many clinicians consider ASPD to be "untreatable", and have largely relegated the management of this challenging disorder to the criminal justice system, effectively relinquishing responsibility for understanding and treating ASPD. Although a number of interventions are utilized by the criminal justice system, these interventions have typically focused on specific problem behaviors, such as anger management and substance abuse. These interventions, along with the more broad-based approaches occasionally studied (e.g., criminal cognitions) focus primarily on cognitive processing, effectively ignoring core elements of ASPD such as impulsivity and emotion dysregulation. Recently, however, growing interest has centered on Dialectical Behavior Therapy as a potential intervention approach, particularly given the emphasis on tangible behaviors and the acquisition of skills to address the core elements of APSD. The proposed study builds upon an innovative rehabilitative program developed by the U.S. District Court in New York. Beginning in 2020, the Fordham Community Mental Health Clinic has provided a DBT-based intervention to participants in this rehabilitation program. This population is comprised of repeat criminal offenders who are deemed at high risk for reoffending by the Probation Department, the vast majority of whom meet diagnostic criteria for ASPD. This intervention, which builds on the researcher team's past work treating offenders with a history of stalking and intimate partner violence, has the potential to advance the utility of DBT for treatment of this challenging population. The present application proposes to advance this goal, by adapting DBT to target core symptoms of ASPD, including impulsivity, difficulties in emotional processing, and problem solving deficits. By adapting traditional DBT, this intervention hopes to demonstrate increased success in retaining and engaging this challenging population in treatment, decreasing the extent of problematic behaviors, and reducing the rates of violent and criminal reoffense. Most importantly, this application takes an experimental therapeutics approach, by identifying potential mediators of successful change in ASPD and quantifying the extent to which DBT impacts these traits and behaviors. Although DBT is not expected to "cure" ASPD, even modest improvements in the treatability of this challenging population would translate into substantial benefits given the high social, economic and health care costs associated with this disorder. Given these goals, the present application seeks to a) demonstrating the feasibility and acceptability of this intervention, b) reduce problematic character traits and behaviors (e.g., decreased impulsivity, increased emotion recognition), and c) reduce the rates of re-offending.

ELIGIBILITY:
Inclusion Criteria:

* Over 18, English speaking, Participating in RISE Court program

Exclusion Criteria:

* Evidence of psychotic symptoms that would preclude meaningful participation in treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criminal offenders on probation in the Southern District of New York's intensive supervision program.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Completion of the treatment program | 4 months after initiation of treatment
  Individuals will be classified as "completers" if they have finished the entire 16 week treatment program

SECONDARY OUTCOMES:
Impulsivitity, | Post-treatment (approximately 4 months after initiation of treatment)
  Impulsivity will be measured with a self-report measure, the UPPS-P Impulsivity Scale, which will be administered prior to, and following completion of treatment
Distress tolerance | Post-treatment (approximately 4 months after initiation of treatment)
  Distress tolerance will be measured with a self-report measure, the Distress Tolerance Scale, which will be administered prior to, and following completion of treatment
Emotion regulation | Post-treatment (approximately 4 months after initiation of treatment)
  Distress tolerance will be measured with a self-report measure, the Difficulties in Emotion Regulation Scale, which will be administered prior to, and following completion of treatment
Mindfulness | Post-treatment (approximately 4 months after initiation of treatment)
  Mindfulness will be measured with a self-report measure, the Mindful Attention Awareness Scale, which will be administered prior to, and following completion of treatment
Renewed criminal charges following completion of treatment | 1 year
  Participants will be monitored for at least one year following treatment in order to determine whether they have been charged with any additional criminal offenses

CONTACTS AND LOCATIONS:
Overall Officials: Barry Rosenfeld, PhD, Principal Investigator — Fordham University
Locations (1):
- Fordham University Community Mental Health Clinic, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Because this is a pilot study it is unclear whether data will be made available to other researchers